CLINICAL TRIAL: NCT05117021
Title: Comparative Study Between Caudal Epidural Block and Ultrasound Guided Transversus Abdominis Plane Block for Post Operative Analgesia in Children Undergoing Infraumblical Surgeries
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Haitham Mohamed Ismail, resident doctor at anesthesia and ICU department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-21-10-40
Record Dates: First submitted 2021-10-17; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Post Operative Analgesia in Children Undergoing Infraumblical Surgeries

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of Bupivacaine injection in Caudal block group (Experimental): The children will receive of 0.25% plain bupivacaine infiltration as caudal block for post operative analgesia in infraumblical surgeries
  Interventions: Drug: Caudal Epidural Block using 0.25% plain bupivacaine dose 1 ml / kg and Ultrasound Guided Transversus Abdominis Plane Block using 0.25% plain bupivacaine dose 0.5 ml / kg
- Group 2 : Group of Bupivacaine injection in TAP block group (Experimental): The children will receive of 0.25% plain bupivacaine infiltration as Transversus Abdominis Plane Block for post operative analgesia in infraumblical surgeries
  Interventions: Drug: Caudal Epidural Block using 0.25% plain bupivacaine dose 1 ml / kg and Ultrasound Guided Transversus Abdominis Plane Block using 0.25% plain bupivacaine dose 0.5 ml / kg

INTERVENTIONS:
Drug: Caudal Epidural Block using 0.25% plain bupivacaine dose 1 ml / kg and Ultrasound Guided Transversus Abdominis Plane Block using 0.25% plain bupivacaine dose 0.5 ml / kg — Caudal Epidural Block and Ultrasound Guided Transversus Abdominis Plane Block using 0.25% plain bupivacaine

SUMMARY:
Comparative study between Caudal Epidural Block and Ultrasound Guided Transversus Abdominis Plane Block for post operative analgesia

DETAILED DESCRIPTION:
Comparative study between Caudal Epidural Block and Ultrasound Guided Transversus Abdominis Plane Block for post operative analgesia in children undergoing infraumblical surgeries

ELIGIBILITY:
Inclusion Criteria:

- 120 children, aged between 4 and 7 years undergoing infraumblical surgeries as ( hypospadias , inguinal hernia and orchopexy ).patients will be selected according to ASA physical status class I to II from both genders who be able to swallow tablets.

Exclusion Criteria:

* parents' refusal.
* urgent cases.
* other contraindications of regional anesthesia (e.g. infection at injection site, coagulopathy and allergy to bupivacaine)
* Insulin dependent diabetes
* Thyroid disease

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
post operative analgesia in infraumblicial surgeries in children children undergoing infraumblical surgeries | 6 months
  Comparative study between Caudal Epidural Block and Ultrasound Guided Transversus Abdominis Plane Block for post operative analgesia in children undergoing infraumblical surgeries.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wang L, Xiao Y, Tian T, Jin L, Lei Y, Finnell RH, Ren A. Corrigendum to "Digenic variants of planar cell polarity genes in human neural tube defect patients." Mol Genet Metab. 2018 May;124(1):94-100. doi:10.1016/j.ymgme.2018.03.005. Epub 2018 Mar 18. https://pubmed.ncbi.nlm.nih.gov/29573971/. Mol Genet Metab. 2021 Mar;132(3):211. doi: 10.1016/j.ymgme.2021.01.010. Epub 2021 Feb 10. No abstract available. PMID 33582009
- [Background] Kumar A, Dogra N, Gupta A, Aggarwal S. Ultrasound-guided transversus abdominis plane block versus caudal block for postoperative analgesia in children undergoing inguinal hernia surgery: A comparative study. J Anaesthesiol Clin Pharmacol. 2020 Apr-Jun;36(2):172-176. doi: 10.4103/joacp.JOACP_100_19. Epub 2020 Jun 15. PMID 33013030
- [Background] Willschke H, Kettner S. Pediatric regional anesthesia: abdominal wall blocks. Paediatr Anaesth. 2012 Jan;22(1):88-92. doi: 10.1111/j.1460-9592.2011.03704.x. Epub 2011 Nov 14. PMID 22077146